CLINICAL TRIAL: NCT07265141
Title: An Automated Virtual Reality Intervention to Enhance Firearm Safety Counseling in Pediatrics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, F. Joseph Real, Associate Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0538; K18HD117377 (NIH)
Record Dates: First submitted 2025-06-13; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality; Medical Education; Motivational Interviewing; Gun Violence Prevention; Artificial Intelligence (AI)
Keywords: virtual reality; Medical Education; Gun violence prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- An Automated Virtual Reality Intervention to Support Firearm Safety Counseling in Clinicians (Experimental): The automated virtual reality intervention allows clinicians to deliberately practice firearm safety counseling skills through verbal interactions with virtual characters with receipt of immediate feedback to support behavior change and mastery learning.
  Interventions: Behavioral: An Automated Virtual Reality Intervention to Support Firearm Safety Counseling in Clinicians

INTERVENTIONS:
Behavioral: An Automated Virtual Reality Intervention to Support Firearm Safety Counseling in Clinicians — The automated virtual reality intervention allows clinicians to deliberately practice firearm safety counseling skills through verbal interactions with virtual characters with receipt of immediate feedback.

SUMMARY:
Clinicians will complete a screen-based automated virtual reality training intervention to learn how to counsel caregivers of pediatric patients on secure firearm storage.

DETAILED DESCRIPTION:
The investigators will recruit pediatric clinicians to participate in an automated screen-based virtual reality intervention. Clinicians will be recruited from clinical locations that offer a variety of setting types (urban, suburban, and rural).

ELIGIBILITY:
Inclusion Criteria:

- Pediatric Clinicians must meet one of the following inclusion criteria at each study site: Physicians (attending, fellow or resident), Licensed Nurse Practitioner, Physician's Assistant

Exclusion Criteria:

* Unable to read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure | From completion of the virtual reality intervention to 2 months
  Four items, Scale score is average across individual items, Minimum score: 1, Maximum score: 5. higher scores indicate better acceptability
Appropriateness of the Intervention Measure | From completion of the virtual reality intervention to 2 months
  Four items, Scale score is average across individual items, Minimum score: 1, Maximum score: 5. higher scores indicate better appropriateness
Feasibility of the Intervention Measure | From completion of the virtual reality intervention to 2 months
  Four items, Scale score is average across individual items, Minimum score: 1, Maximum score: 5. higher scores indicate better feasibility

SECONDARY OUTCOMES:
De Novo Survey Item for Assessing Social Cognitive Theory Construct Behavioral Capability | From completion of the virtual reality intervention to 2 months
  One item, Scale score of individual items, Minimum score: 1, Maximum score: 5. higher score indicates more behavioral capability
De Novo Survey Items for Assessing Social Cognitive Theory Construct Self-Efficacy | From completion of the virtual reality intervention to 2 months
  Eight items, Scale score for individual items, Minimum score: 0, Maximum score: 4. Higher scores indicate more self-efficacy.
De Novo Survey Items for Assessing Social Cognitive Theory Construct Expectations | From completion of the virtual reality intervention to 2 months
  Three items, Scale score of individual items, Minimum score: 1, Maximum score: 5. Higher scores indicate more expectations.
De Novo Survey Items for Assessing Social Cognitive Theory Construct Expectancies | From completion of the virtual reality intervention to 2 months
  Six items, Scale score of individual items, Minimum score: 1, Maximum score: 5. higher scores indicate higher expectancies for prioritizing firearm safety discussions across different ages for well-child visits.

OTHER OUTCOMES:
De Novo Standardized Patient Encounter Assessment Tool - Assessing Fidelity to the Virtual Reality Intervention Components | From completion of the virtual reality intervention to 6 months
  Participant's will engage in a standardized patient encounter to assess fidelity to behavioral skills reviewed during the virtual reality intervention, 20 items, maximum score: 20, minimum score: 0, scaled scores for firearm counseling skills and motivational interviewing skills, scaled scores determined by adding together individual items, 17 items related to firearm safety counseling, 3 items related to motivational interviewing

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) for survey data will include clinician participants' (a maximum of n=30) demographic data (race, age, gender, role, practice setting, experience counseling on firearm safety), responses to items related to implementation (acceptability, appropriateness, and feasibility), and responses to items related to psychosocial constructs (behavioral capability, self-efficacy, expectations and expectancies). Data will include demographic information, baseline characteristics, outcome measures, and adverse event data. Access will be granted to researchers with a methodologically sound proposal, subject to review by the study team and institutional policies. Data be to be shared will be archived in DASH through the NICHD repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data access included in associated publications or the end of the award period, whichever comes first.
Access Criteria: Requests for data access should be submitted to the Principal Investigator or through the data sharing plan website.
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Background] March M, Zackoff M, Fleck J, Meisman A, Humphrey K, MacDougall MC, Ehrlich S, Griggs C, Sacks C, Masiakos P, Klein M, Real F. A Randomized Trial of Virtual Reality Training to Improve Firearm Safety Counseling Skills. Acad Pediatr. 2025 Jan-Feb;25(1):102560. doi: 10.1016/j.acap.2024.08.005. Epub 2024 Aug 10. PMID 39128562
- [Background] Real FJ, Griggs C, March M, Masiakos PT, Meisman A, Felopulos G, Sacks CA, Zackoff MW. Feasibility and Acceptability of a Virtual Reality Curriculum to Support Firearm Safety Counseling Skills Among Pediatric Residents. J Grad Med Educ. 2024 Dec;16(6):740-746. doi: 10.4300/JGME-D-24-00022.1. Epub 2024 Dec 13. PMID 39677314
- [Background] March ML, Meisman AR, Zackoff MW, Klein MD, Real FJ. Caregivers' and Community Members' Perspectives on Firearm Safety Screening and Counseling During Pediatric Primary Care Visits. J Pediatr Clin Pract. 2024 Mar 14;12:200099. doi: 10.1016/j.jpedcp.2024.200099. eCollection 2024 Jun. PMID 39949418